CLINICAL TRIAL: NCT05364892
Title: Biocollection of Patients With ANCA Associated Vasculitis Diagnosed Within the CERAINO Autoimmune Disease Reference Center, Part of the Global BRAISE Project (B-dependent Rare AutoImmune DiseaSES
Brief Title: Biocollection of Patients With ANCA Associated Vasculitis
Acronym: ANCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC20.0233
Record Dates: First submitted 2020-12-21; First posted 2022-05-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-01

CONDITIONS: ANCA-associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Diagnosis and follow up of ANCA-associated vasculitis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANCA-associated vasculitis - patient library (Other): It is a description of ANCA-associated vasculitis patients cohort. All the patients are included in one arm. They will undergo various type of samples.
  Interventions: Other: Blood samples (80 mL); Other: Fecal samples; Other: Urinary sample (20-40 mL); Other: Questionnaires

INTERVENTIONS:
Other: Blood samples (80 mL) — Blood samples (80 mL) at inclusion, once a year for 5 years, and if relapse or change of treatment
Other: Fecal samples — Fecal samples at inclusion
Other: Urinary sample (20-40 mL) — Urinary samples at inclusion, once a year for 5 years, and if relapse or change of treatment
Other: Questionnaires — Questionnaires at inclusion, once a year for 5 years, and if relapse or change of treatment

SUMMARY:
As rare disease, vasculitis affects a small number of patients, the cohorts available in the literature are few and the pathophysiological mechanisms remain to be elucidated. The collection of standardized data within a patientheque as part of a multi-year follow-up will facilitate the study of the characteristics of these diseases. This may, in particular, address the main objective of identifying predictors of relapse, as well as secondary objectives for predictive factors of mortality, infectious, cardiovascular or neoplastic complications that affect the prognosis of vasculitis in order to establish a more appropriate management of the patients concerned.

DETAILED DESCRIPTION:
Vasculitis associated with anti-neutrophil cytoplasm antibodies (ANCA) is a group of rare and severe autoimmune diseases, encompassing several entities: granulomatosis with polyangiitis (GPA), microscopic polyangiitis (PMA), and eosinophilic granulomatosis with polyangiitis (GEPA). When untreated, these diseases are fatal in a matter of months. Currently, thanks to the use of corticosteroids and immunosuppressants, this high mortality has greatly decreased and these are now chronic diseases. On the other hand, these patients are at high risk of morbidity, linked to both relapses (occurring in at least 50% of patients) and side effects of treatments. It is therefore essential to be able to define which patients are at risk of relapse and justify long-term immunosuppressive treatment to avoid recurrence of the disease, and conversely which patients have a low risk of relapse and in whom immunosuppressive treatments can be discontinued to limit the risk of side effects. However, so far no predictor or biomarker can accurately assess this risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with no upper age limit.
* Patients assessed as part of the reference centre for rare autoimmune diseases at the CHRU in Brest.
* Patients for whom a diagnosis of ANCA-associated vasculitis is made by the physician in charge of the patient, according to the definitions of the Chapel-Hill Consensus Conference.
* Patient affiliated with Social Security
* Patient who has signed written informed consent

Exclusion Criteria:

* Minor
* Patients unable to consent.
* Patients refusing to participate in research
* Patient under legal protection (tutelage, curatorship)
* Pregnant or lactating women
* Hemoglobin (Hb) < 7g/dL

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2032-10-27 (Estimated); Study Completion 2032-10-27 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival of the disease | Five years after diagnosis
  Relapse-free survival of the disease

SECONDARY OUTCOMES:
death | Five years after diagnosis
  death
Age | Five years after diagnosis
  Age
Sex | Five years after diagnosis
  Sex
Physician assessment of disease activity | Five years after diagnosis
  Disease activity will be assessed on a scale from 0 to 100, considering the pain and the impact on daily life. A higher score means a worse outcome.
Patient assessment of disease activity | Five years after diagnosis
  Disease activity will be assessed on a scale from 0 to 100, considering the pain and the impact on daily life. A higher score means a worse outcome.
BVAS score - Birmingham Vasculitis Activity Score | Five years after diagnosis
  Questionnaire listing 56 symptoms divided into nine organ/systems classes, plus an "other" section. For each item, the assessor evaluates if it is present and attribuable to the active vasculitis or not. A higher score means a worse outcome.
VDI score - Vasculitis Damage Index | Five years after diagnosis
  This is for recording organ damage that has occurred in patients since the onset of vasculitis, and over 3 months. Record features of active disease using the Birmingham Vasculitis Activity Score (BVAS).
  A new patient should usually have a VDI score of zero, unless:
  1. they have had vasculitis for more than three months of onset of disease. and
  2. the damage has developed or become worse since the onset of vasculitis Questionnaire listing 64 symptoms divided into eleven organ/systems classes. For each item, the assessor evaluates if it is present over 3 months and attribuable to the active vasculitis or not. A higher score means a worse outcome.
Number of patients with refractory character of the Vasculitis | Five years after diagnosis
  Number of patients for whome a secondary decision to intensify immunosupressive treatment in the first year of treatment (increased corticosteroid dosage, introduction of another immunosupressor outside the scheduled at the end of the initial assessment) has been taken.
HAQ-DI - Health Assessment Questionnaire - Disability Index. | Five years after diagnosis
  Evolution of HAQ-DI during follow-up 8 fields questionnaire (DRESSING & GROOMING, ARISING, EATING, WALKING, HYGENE, REACH, GRIP, Other activites), scaled from 0 to 3, 3 meaning a worse outcome.
Glucocorticoid toxicity index - Glucocorticoid toxicity index during follow-up Glucocorticoid toxicity index | Five years after diagnosis
  Glucocorticoid toxicity index during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest - Service de rhumatologie, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement